CLINICAL TRIAL: NCT05244317
Title: Removable Splint Versus Cast in the Treatment of Distal Radius Fracture in Children of Refugees' Camps: a Randomized Controlled Trial
Brief Title: Removable Splint Versus Cast in the Treatment of Distal Radius Fracture in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no cases included
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Jagar Omar Doski, Assistant Professor of Orthopedics, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDuhok
Record Dates: First submitted 2022-01-15; First posted 2022-02-17 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Fracture of Radius
Keywords: splint; cast
MeSH Terms: conditions — Radius Fractures | interventions — Casts, Surgical; Splints

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cast group (Placebo Comparator): treatment of the participant of this group will be by the standard method which is by casting
  Interventions: Device: cast
- splint group (Experimental): treatment of the participant of this group will be by the removable splint
  Interventions: Device: splint

INTERVENTIONS:
Device: cast — the cast of the upper limb from just below elbow joint to the knuckle of fingers
  Arms: cast group
Device: splint — Removable splint
  Arms: splint group

SUMMARY:
Refugees live in camps under unusual living conditions. The children in the camps may not have enough safe facilities to play. If an injury occurred in these children, the classical and adequate regime of treatment may not be available. Hence, it may be valuable to find simple, cheap, and safe methods of treatment for their injuries.

DETAILED DESCRIPTION:
Fractures of the distal forearm (especially radius) are the most common fracture reported in childhood and a frequent reason for visiting the emergency unit and orthopedic clinic in hospitals. Because of the age of patients and proximity to the joint, these fractures heal well and have a good ability to remodel the bone even with mild displacement. Therefore, most of these fractures are treated conservatively by a short arm cast with frequent visits to the orthopedic clinic within 4-6 weeks without significant complications. Several studies report successful treatment of these fractures by removable splint as a substitute for the cast. The splints proved to be safe and cost-effective in managing these common minor injuries in children under usual living conditions.

Refugees live in camps under unusual living conditions. The children in these camps may not have enough safe facilities to play. If they got an injury, the classical and adequate regime of treatment may not be available. Hence, it may be valuable to find simple, cheap, and safe methods of treatment for their injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 2-12 years old age.
* Sex: both male and female.
* Address: living in one of the refugees' camps in the Duhok Government.
* Duration of symptoms: less than 7 days.
* Type of injury: fracture at the distal end of radius proofed by a radiograph film in two views (posteroanterior and lateral).
* Type of fracture: it may be any of the followings:

  * torus (buckle) fracture,
  * undisplaced or minimally displaced fracture distal radius physis (type 1 and 2 only) that do not need reduction.
  * undisplaced or minimal displaced metaphyseal fracture that does not need reduction. Note: The minimally displaced fracture will be considered when the fracture fragments have a tilt of fewer than 15 degrees and shift less than 5 millimeters at the fracture site in both views.

Exclusion Criteria:

* open fractures
* pathological fractures
* displaced fractures that need reduction
* delayed presentation beyond 7 days
* associated fracture of the ulnar bone
* polytraumatic cases.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
complication | up to 12 weeks.
  proportion of complication occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jagar O Doski, Study Chair — University of Duhok
Locations (1):
- Jagar Omar Doski, Duhok, Duhok Governorate / Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
personal contact with the investigator